CLINICAL TRIAL: NCT05969535
Title: The Effect of Education Given Accordıng to the Travelbee Human Human Relatıons Model On Prenatal Attachment, Birth Fear and Anxiety in Pregnants With Fear of Birth
Brief Title: The Effect of Education Given to Pregnancy on Prenatal Attachment, Anxiety and Fear of Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuğba Sarı (Other)
Responsible Party: Sponsor-Investigator, Tuğba Sarı, Sponsor Investigator, Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: TOGU-HEM-TS-01
Record Dates: First submitted 2023-07-12; First posted 2023-08-01 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Fear of Childbirth
Keywords: fear of childbirth; prenatal attachment; anxiety; pregnancy; human to human relationship
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: According to the WIJMA version A scale, two groups will be formed by randomization method as intervention and control group for pregnant women who are determined to have fear of middle and higher birth. 8 sessions of psychoeducation program will be given to the pregnant women in the intervention group. The control group will continue routine monitoring. After the training, the level of fear of birth, prenatal attachment and anxiety levels will be compared between the two groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): This group will consist of 35 primiparous pregnant women. The training program, prepared in line with travelbe's human-human relations model, will continue for a total of 4 weeks, 2 days a week.
  Interventions: Behavioral: Birth preparation education according to travelbee human-human relations theory
- control group (No Intervention): This group will consist of 35 primiparous pregnant women. No training program will be given to this group and routine pregnant follow-up will continue.

INTERVENTIONS:
Behavioral: Birth preparation education according to travelbee human-human relations theory — human-to-human communication and psychoeducation-assisted birth preparation training
  Arms: intervention group

SUMMARY:
Communication between nurse and patient is considered essential to provide holistic and humane care as it allows patients to be fully understood, assisted, and their needs defined as empathetic. Travelbee, states that nursing is conducted through human-to-human relationships. These relationships begin first with the encounter of the nurse and the patient, then with the stage of emergence of identities where the relationship begins, the stage in which the nurse and the patient perceive each other's uniqueness, the empathy stage in which the person shares their experiences, the sympathy stage in which the nurse wants to reduce the cause of the patient's pain, and the final stage is the nurse and the patient's interrelated thoughts and feelings, their interest and concern towards others, a non-judgmental attitude and a person specific to each individual it consists of the stage of harmony that he approaches with respect. During this biological process, many physiological and psychological changes can be expected in pregnant women. Many psychological and social factors influence the fear of childbirth. These factors include; Lack of self-confidence in childbirth, being affected by negative birth histories, history of depression, anxiety, partner dissatisfaction, young maternal age, low income level, low education and low perception of social support, pain in childbirth or fear of losing control, and physical injury during childbirth. It is also possible that the fear of childbirth and the appearance of symptoms of stress and anxiety, which complicates pregnancy. Mother-infant bonding, which is adversely affected by mental problems such as anxiety, depression and fear of childbirth during pregnancy, can adversely affect the attachment process in both prenatal period. There are some non-pharmaceutical applications to strengthen the mental health of the mother, to reduce stress and fear of childbirth, and to strengthen the mother-baby bond. These are practices that include listening to music, psychoeducation, cognitive and behavioral therapies. With professional support in this study, childbirth will take place in a completely safe environment where stress and fear of childbirth are less. Nurses need to communicate from person to person in order to achieve the goal of effective care and to be healing. The training program was created based on Travelbee's five-step human-to-human relationship model with pregnant women who fear childbirth.

DETAILED DESCRIPTION:
Type of Research The research will be conducted as a randomized controlled treatment study aimed at directing the education given according to the Travelbee human explanation theory to the fear of birth, prenatal retention and anxiety in primiparous pregnant women who have fear of childbirth.

The Universe of the Research The population of the research consists of primiparous pregnant women who came to the Obstetrics and Gynecology outpatient clinic between July 2023 and October 2023.

Sample of the Research G*Power version 3.1.9.7 program was used to calculate the size and power value of the research sample. It was calculated by taking a reference to a study done in the sample size calculation. According to the G power analysis, 5% margin of error, 95% power (representing the universe) and an effect size of 1.031 were calculated as 26 in total, 52 in both groups. As the main parameter of the study in the selection of the sample, the pregnant women with moderate and high level of fear of childbirth score from the Wijma Birth Expectation / Experience Scale (W-DEQ) Version A scale will be selected. In the literature review, the fear of childbirth starts from the 20th week of pregnancy and increases during pregnancy. Therefore, pregnant women with 20th gestational week and older than this week were included in the study. In order for the training program to be 4 weeks and for the participating pregnant women to complete prenatal education, pregnant women after 34 weeks were not included. Considering the loss of pregnant women who met the research criteria and accepted to participate in the study, the sample size was determined as 70 participants, 35 for both groups.

Formation of the Control and Experimental Group After meeting the pregnant women who came for the routine pregnancy examination and evaluating whether it was the first pregnancy according to the research criteria, the Personal Information Form and the Wijma Birth Expectation / Experience Scale Version A scale were filled out by the pregnant women who met the inclusion criteria. Pregnant women with a medium or higher fear of childbirth score were informed about the study and their verbal and written consent was obtained from the voluntary consent form. In addition, a list has been prepared including the name and surname of the pregnant women, the estimated date of birth according to the last menstrual period, and contact information.

Randomization Randomization technique was used to assign participants to groups. The stratification randomization technique will be used to ensure homogeneity according to the data obtained from the pregnant women (educational status, age and fear of childbirth).

Blinding It is not suitable for double blinding because the researcher included in the study provided education according to Travelbee human-human relations theory, collected data on fear of birth, prenatal attachment and anxiety, and took part in the analysis of these data. However, because the pregnant women were assigned to the experimental and control groups by randomization method and the individuals did not interact with each other and did not know which group they were in, unilateral blinding would be applied.

Variables of the Study Dependent variables: prenatal attachment inventory total score, wijma birth expectancy/experience scale version A score, beck anxiety scale total score.

Independent variables: Psychoeducation prepared according to Travelbee human-human relations model within the scope of the study.

Control variables: Age, income and education level, employment and social security status, family type, region of residence, gestational week, age at marriage and obstetric characteristics of pregnant women constitute control variables.

Application of Research The research was carried out within the framework of three separate stages. Phase 1: Preparation phase "Travelbee Human-Human Relations Theory-Based Training Program for Reducing Fear of Birth" at the preparatory stage "Birth Preparation Training" guide has been developed. Stage 2: Pre-implementation stage of the training program Stage 3: Implementation stage of the training program

Preparation Process of the Training Program Within the scope of the training program, the studies and training contents were examined in order to help women with their first pregnancy cope with the fear of childbirth, to determine the negative emotional state caused by the fear of birth and to reduce its effects, and to increase prenatal attachment, and a training plan was created in this direction. The educational content of the study was created in line with the five steps (acquaintance, emergence of identities, empathy, sympathy, adaptation stage) of the Travelbee human-human relations model. While these steps were being created, psychoeducational approaches were examined in line with the literature, and the techniques of making people aware of dysfunctional thoughts, asking questions, recognizing automatic thoughts, giving homework and feedback techniques were used in the training content. Opinions were received from 7 experts from the field of mental health and diseases nursing and one expert in the field of psychiatry regarding the training content created.

Purpose of the Prepared Training Program The training program aims to realize the fear of childbirth and the negative emotional state caused by this fear in women experiencing their first pregnancy within the scope of preparation for childbirth and to help them cope with it, to make them realize the importance of prenatal attachment and to increase attachment. The main subjects of the training content given to the pregnant women who participated in the training during the group process;

* Defining and evaluating pregnancy and birth perception
* The importance of childbirth preparation classes
* Evaluation of fear of childbirth and anxiety
* Evaluation of beliefs and attitudes towards birth
* Evaluation of fear of childbirth and its normalization and individual reactions
* The stage of preparation for birth and the importance of prenatal attachment
* Evaluation of the existence of fear of childbirth and normalization social supports
* Evaluation of communication and cooperation in baby care

Pre-application Pre-application, training program was started with 15 primiparous pregnant women, but they were excluded from the study because one pregnant had transportation problems and two pregnants found the education period long and wanted to withdraw from the study. Pre-application was made with 12 primiparous pregnant women. In order to evaluate the duration of the training, its intelligibility, the appropriateness of the subjects and its effect on the fear of childbirth, and the subjects that can be changed, the training was applied twice a week for 4 weeks. With the pre-application, no changes were made in the subjects, but changes were made in the predetermined training periods. Pregnant women who were included in the preliminary application were not included in the experimental and control groups of the study.

Implementation of the Experimental Group Training Program Within the scope of the research, the suitability of the place, time and hour of the training will be determined by interviewing the primiparous pregnant women in the experimental group. After discussing with all pregnant women and determining the appropriate time and day for everyone, the days when there are no trainings will be planned in the pregnant training school of the hospital. Travelbee Human-Human Relations Theory-Based Training Program for Reducing Birth Fear and Anxiety and Increasing Prenatal Attachment A training program of eight sessions will be applied to pregnant women between 20th and 34th weeks, twice a week for four weeks.

Session 1 First Encounter Phase (Introduction) Session 2 Revealing Identities (Group Members Getting to Know Each Other and Awareness of the Group's Purpose) Session 3 Empathy Stage (Recognition and Evaluation of Birth Action, Evaluation of Misinformation, Beliefs and Attitudes towards Birth) Session 4 Empathy Phase (Defining and Evaluating Fear of Birth) Session 5 Sympathy Phase (Coping with Birth Contractions) Session 6 Sympathy Stage (The Importance of Birth Preparation and Prenatal Attachment) Session 7 Adjustment Phase (Pregnancy Process and Presence of Social Supports, Evaluation of Baby Care) Session 8 Evaluation (Group Feedback and Termination)

Control Group Within the scope of the research, no intervention will be made to the pregnant women in the control group between the 20th and 34th weeks, apart from the routine hospital practices.

Collection of Research Data After the data were met with the pregnant women who came to the obstetrics and gynecology outpatient clinic before or after their outpatient clinic examinations and were informed about the research, the introductory information form and the Wijma birth expectation / experience scale version A were filled by the pregnant women who accepted the study. From this scale, the pregnant women who accepted the study were selected among the pregnant women with a medium or higher fear of childbirth score. Contact information was obtained from the accepted pregnant women. Experimental control groups were formed by stratified randomization to ensure within-group homogeneity, and the Prenatal Attachment Inventory and Beck Anxiety Scale, which are pretest data collection tools, will be filled in the first session. In the training program prepared within the scope of the research, the intervention will be applied to the pregnants in the experimental group, in the form of eight sessions in total, at least once a week, at most two sessions, while the control group will continue their routine follow-up. After the training program is completed, Prenatal Attachment Inventory, Wijma Birth Expectation/Experience Scale Version A, Beck Anxiety Scale will be administered again in the last session to obtain post-test data. In order to ensure homogeneity and to use the time appropriately, the pregnant women in the experimental group will be divided into three groups.

Analysis of Research Data The descriptive statistics for the quantitative variables of the research determined by measurement will be shown as mean and standard deviation and percentage. First of all, the conformity of the data to the normal distribution will be evaluated with the Shapiro-Wilk test. In the analysis of normally distributed data as a result of the Shapiro-Wilk test, ANOVA between three or more variables and t-test in independent groups in pairwise comparisons, Mann-Whitney U test in pairwise comparisons between two-category variables in the analysis of non-parametric data, and Kruskal-Wallis H-test in order to find the differences between variables with three or more categories. Correlation analysis will be performed to reveal the relationship between dependent variables. In addition, Wilcoxon test (significance test of difference between two spouses) will be used to test the difference in two different measurement times obtained from the same individuals. The difference between categorical variables will be evaluated with the Pearson chi-square test. A value of 0.05 will be accepted as the level of significance in the entire study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over.
* At least primary school graduate.
* According to the last menstrual period or for pregnant women who do not know the last menstruation date, to be between 20-34 weeks in the calculations made with USG data.
* Intermediate and higher score on the Wijma birth expectancy/experience scale version A.
* Having a single and live pregnancy.
* Having your first pregnancy.
* Agreeing to participate in the research.
* Having trouble communicating.
* No infertility treatment.
* No contraindications for vaginal delivery

Exclusion Criteria:

* Pregnant women with medical indications.
* Those with high-risk pregnancies.
* Having given birth before.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Since there is a training program on pregnant women, female gender was preferred.
Enrollment: 62 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Wijma Birth Expectation/Experience Scale (W-DEQ) Version A | each participant pregnant will be evaluated for outcome measure for four weeks
  It is a scale developed to determine the birth fear and stress of pregnant women. W-DEQ version A is a 6-point Likert-type scale consisting of 33 items. While the minimum score on the scale is 0, the maximum score is 165. The negatively charged questions (2, 3, 6, 7, 8, 11, 12, 15, 19, 20, 24, 25, 27, 31) in the scale are calculated by reversing them. A high score indicates a high level of fear of childbirth. The cutoff point is 85. A score of 85 and above indicates clinical fear of childbirth. The Cronbach's Alpha value of the scale was found to be 0.88 for primiparous pregnants and 0.90 for multiparous pregnants.
  * 0-37 points = mild fear of childbirth
  * 38-65 points = moderate fear of childbirth
  * 66-84 points = severe fear of childbirth
  * 85 and above = clinical fear of childbirth
Beck Anxiety Scale (BAI) | each participant pregnant will be evaluated for outcome measure for four weeks
  It is a scale developed to measure anxiety symptoms and reveal the cognitive aspects of anxiety. The scale consists of 21 items and is a four-point Likert type scale scored between 0-3. The lowest 0 and the highest 63 points are obtained in the scale. For each item, it is required to tick one of the options "None", "Mild", "Moderate", "Severe". 13 items evaluate physiological symptoms, 5 items describe the cognitive aspect, 3 items represent both somatic and cognitive symptoms. The high total score obtained in the scale indicates the severity of the anxiety experienced by the individual. The Cronbach alpha value of the scale was found to be 0.93.
Prenatal Attachment Inventory (PAI) | each participant pregnant will be evaluated for outcome measure for four weeks
  Prenatal attachment inventory was developed to explain the thoughts, feelings and experiences of pregnant women and to determine mother-baby attachment levels. The scale is applied to pregnant women in the 20th and 40th weeks of pregnancy. The scale consists of 21 items. A minimum of 21 points and a maximum of 84 points can be obtained from the scale. An increase in the score indicates that the level of attachment to the baby also increases. The Cronbach Alpha reliability coefficient of the scale was stated as 0.84.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Sarı, Nurse, Principal Investigator — Yozgat City Hospital
Locations (1):
- Yozgat City Hospital, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected and affecting the outcome of the study will be published
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication
Access Criteria: Only the collected data will be shared for analysis.